CLINICAL TRIAL: NCT00912145
Title: Bioavailability of Alprazolam Tablets, 2 mg.
Brief Title: To Demonstrate the Relative Bioavailability of Alprazolam Tablets, 2 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 005-35-11034
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-06

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Alprazolam

ARMS (2):
- 1 (Experimental): Alprazolam Tablets, 2 mg (Geneva Pharmaceuticals, Inc.)
  Interventions: Drug: Alprazolam Tablets, 2 mg (Geneva Pharmaceuticals, Inc.)
- 2 (Active Comparator): Alprazolam Tablets, 2 mg, Xanax (The Upjohn Company)
  Interventions: Drug: Alprazolam Tablets, 2 mg (Geneva Pharmaceuticals, Inc.)

INTERVENTIONS:
Drug: Alprazolam Tablets, 2 mg (Geneva Pharmaceuticals, Inc.)

SUMMARY:
To Demonstrate the Relative Bioavailability of Alprazolam Tablets, 2 mg.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 19 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 1996-02; Primary Completion 1996-02 (Actual); Study Completion 1996-02 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 13 days

CONTACTS AND LOCATIONS:
Overall Officials: Calvin F. Fuhrmann, M.D., Principal Investigator — PharmaKinetics Laboratories Inc.